CLINICAL TRIAL: NCT03671551
Title: Study of Psychomotor Development and Attachment in Children Aged 6 to 30 Months With Oral Disorder
Acronym: TODEVA
Status: Terminated | Type: Observational
Why Stopped: Recruitment too low
Sponsor: Camille JUNG (Other)
Responsible Party: Sponsor-Investigator, Camille JUNG, Head of the clinical research department, Centre Hospitalier Intercommunal Creteil
Organization: Centre Hospitalier Intercommunal Creteil (Other)
Other Study IDs: TODEVA
Record Dates: First submitted 2018-08-08; First posted 2018-09-14 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Eating Disorders in Children; Psychomotor Development Impaired
Keywords: Eating Disorders in Children; Psychomotor Development Impaired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psychomotor/psychological evaluation: Children in the study aged 6 to 30 months followed or referred to CHIC for oral disorders will have a psychomotor assessment and a psychological interview. Questionnaires on eating behavior will also be proposed.

SUMMARY:
Dietary difficulties and eating disorders of the child are a common reason for consulting infants and young children. There is currently little data on the psychomotor development of these children and their association with parent-child attachment. The objective of this study is to evaluate, at the same time, the three physiological, psychomotor and attachment dimensions of children with eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 to 30 months
* Oral disorder defined by a MCH score ≥ 61

Exclusion Criteria:

* Children in enteral nutrition asked for an indication other than oral disorders
* Children followed for serious chronic organic pathology causing disorders of the oral (DNTC, swallowing disorders, etc.)
* Child already assessed by the psychomotrician who participated in the study
* Placement of the child in a medical institution or in a foster family.
* Parents' refusal to participate in the study
* Establishment of a psychomotor follow-up between the time of the medical consultation and the psychomotor evaluation.

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged from 6 to 30 months with eating disorder and adressed by the pediatrician or general practitionner
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Developmental Quotient | at day 1
  Developmental Quotient at Brunet Lézine revised

SECONDARY OUTCOMES:
Quotient of development of the posturo-motor skills | 1 day
  Quotient of development of the posturo-motor subcategory with revised Brunet Lézine
Development Quotient for the Brunet Lézine Coordination Subcategory | 1 day
  Development Quotient for the Brunet Lézine Coordination Subcategory
Developmental Quotient for Brunet Lézine Language Subcategory | 1 day
  Developmental Quotient for Brunet Lézine Language Subcategory
Development Quotient for the Brunet Lézine Socialization Subcategory | 1 day
  Development Quotient for the Brunet Lézine Socialization Subcategory
tactile irritability | 1 day
  Rating on the evaluation grid with tactile irritability
irritant irritability | 1 day
  Scorecard score at irritant irritability
Observation of attachment | 1 day
  Score at the grid observation of attachment lines before, during and after the separation of the child
Attachment with grandparent / parent | 1 day
  Terms of Description of Grandparent / Parent and Parent / Child Attachment by Qualitative Analysis to Semi-directed Issues on Attachment
Food difficulty score child eating behavior questionnaire | 1 day
  Food difficulty score child eating behavior questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Camille JUNG, MD, Principal Investigator — CHI Créteil
Locations (2):
- France (2):
  - CHI Creteil, Créteil
  - CHI Créteil, Créteil, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammaniti M, Lucarelli L, Cimino S, D'Olimpio F, Chatoor I. Feeding disorders of infancy: a longitudinal study to middle childhood. Int J Eat Disord. 2012 Mar;45(2):272-80. doi: 10.1002/eat.20925. Epub 2011 Apr 14. PMID 21495054
- [Background] Cardona Cano S, Tiemeier H, Van Hoeken D, Tharner A, Jaddoe VW, Hofman A, Verhulst FC, Hoek HW. Trajectories of picky eating during childhood: A general population study. Int J Eat Disord. 2015 Sep;48(6):570-9. doi: 10.1002/eat.22384. Epub 2015 Jan 30. PMID 25644130
- [Background] Dubedout S, Cascales T, Mas E, Bion A, Vignes M, Raynaud JP, Olives JP. [Feeding disorders in infants and toddlers: At-risk situations and predisposing factors]. Arch Pediatr. 2016 Jun;23(6):570-6. doi: 10.1016/j.arcped.2016.03.015. Epub 2016 Apr 25. French. PMID 27133367
- [Background] Kerzner B, Milano K, MacLean WC Jr, Berall G, Stuart S, Chatoor I. A practical approach to classifying and managing feeding difficulties. Pediatrics. 2015 Feb;135(2):344-53. doi: 10.1542/peds.2014-1630. Epub 2015 Jan 5. PMID 25560449
- [Background] Le Heuzey MF. [Child food refusal: when will we call a child psychiatrist?]. Arch Pediatr. 2011 Aug;18(8):917-20. doi: 10.1016/j.arcped.2011.05.014. Epub 2011 Jun 16. French. PMID 21683562
- [Background] Issanchou S, Nicklaus S. [Early determinants of food behaviour]. Arch Pediatr. 2010 Jun;17(6):713-4. doi: 10.1016/S0929-693X(10)70073-7. No abstract available. French. PMID 20654855
- [Background] Quah PL, Chan YH, Aris IM, Pang WW, Toh JY, Tint MT, Broekman BF, Saw SM, Kwek K, Godfrey KM, Gluckman PD, Chong YS, Meaney MJ, Yap FK, van Dam RM, Lee YS, Chong MF; GUSTO Study Group. Prospective associations of appetitive traits at 3 and 12 months of age with body mass index and weight gain in the first 2 years of life. BMC Pediatr. 2015 Oct 12;15:153. doi: 10.1186/s12887-015-0467-8. PMID 26459321